CLINICAL TRIAL: NCT02287090
Title: Comparative Effectiveness of Operative Versus Non-Operative Treatments for Rotator Cuff Tears
Acronym: ROW
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Brigham and Women's Hospital (Other); Orthopedic Institute, Sioux Falls, SD (Other); University of Texas (Other)
Responsible Party: Principal Investigator, Nitin Jain, Associate Professor of Physical Medicine and Rehabilitation and Orthopaedics, Vanderbilt University
Other Study IDs: 140857; K23AR059199 (NIH)
Record Dates: First submitted 2014-11-03; First posted 2014-11-10 (Estimated); Last update posted 2025-02-06 (Actual); Status verified 2024-10

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Observational Cohort

SUMMARY:
Rotator cuff tears are one of the most common causes of shoulder pain. Evidence-based guidance on optimal diagnostic and treatment strategies for rotator cuff tears is lacking. Our proposed study aims to fill these gaps by identifying the prognostic factors which will predict better outcomes of rotator cuff tears, based on both operative and non-operative treatment. The investigators will also compare outcomes of operative and non-operative treatment of rotator cuff tears and report on the best way to diagnose rotator cuff tears.

DETAILED DESCRIPTION:
Rotator cuff tears account for over one quarter million surgeries annually. They are a leading cause of shoulder pain and disability. Patients with rotator cuff tears present with shoulder pain and/or limitation in range of motion. Fourteen special physical exam tests have been described for diagnosis of rotator cuff tears. Prior literature describing sensitivity and specificity of these tests in diagnosing cuff tears is limited by retrospective design, small sample sizes, samples restricted to patients undergoing surgery, and failure to differentiate between partial and full thickness tears. As a result, there is little evidence to help clinicians interpret the diagnostic value of the clinical exam. Consequently, clinicians rely heavily on magnetic resonance imaging (MRI) for diagnosing cuff tears, adding considerable expense in the diagnostic process.

The treatment options for rotator cuff tears are operative and non-operative. There is currently little consensus on indications and timing of rotator cuff surgery or non-operative treatment. Furthermore, there is lack of evidence-based guidance on factors associated with outcomes of operative versus non-operative treatment for cuff tears.

We are enrolling patients in a prospective cohort study to assess comparative-effectiveness of operative versus non-operative treatment of rotator cuff tears and understand prognostic factors for better outcomes after surgery and non-operative treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 or older
* Symptoms for at least 4 weeks of shoulder pain and/or limitation in range of motion of shoulder

Exclusion Criteria:

* History of humeral fractures
* Prior surgery on the same shoulder
* Contraindications to MRI (prior surgical hardware, pacemakers, defibrillators, and claustrophobia)
* Unable or unwilling to give informed consent
* Unable or unwilling to be followed up
* Non-English speaking (as questionnaires have only been validated in English)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the clinic with rotator cuff tears.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2011-03 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2024-12 (Actual)

PRIMARY OUTCOMES:
Pain/Function (as measured by the SPADI outcome score) | 24 months
  Comparing patient pain/function [as measured by the Shoulder Pain and Disability Index (SPADI) outcome instrument] between patients undergoing surgery and patients choosing non-operative treatment.

SECONDARY OUTCOMES:
Pain/Function (as measured by the ASES outcome score) | 24 months
  Comparing patient pain/function [as measured by the American Shoulder and Elbow Society (ASES) outcome instrument] between patients undergoing surgery and patients choosing non-operative treatment.
Pain/Function (as measured by the QuickDash outcome score) | 24 months
  Comparing patient pain/function [as measured by the Disabilities of the Arm, Shoulder and Hand (QuickDASH) score] between patients undergoing surgery and patients choosing non-operative treatment.
Effects of rotator cuff tear size on outcomes (as measured by the SPADI outcome instrument). | 24 months
  To determine the effect of rotator cuff size tear (as measured by MRI) on outcome [as measured by the Shoulder Pain and Disability Index (SPADI) outcome instrument], controlling for surgical/non-operative treatment.
Effects of patient age on outcomes (as measured by the SPADI outcome instrument). | 24 months
  To determine if patient age affects their outcome [as measured by the Shoulder Pain and Disability Index (SPADI) outcome instrument], controlling for surgical/non-operative treatment.

OTHER OUTCOMES:
Sensitivity/specificity of symptoms and physical exam (compared with MRI and expert clinicians' diagnosis) | 24 months
  To determine the sensitivity/specificity of symptoms and physical examination as compared with MRI and expert clinicians' diagnosis for the detection of rotator cuff tears.

CONTACTS AND LOCATIONS:
Overall Officials: Nitin B Jain, MD, MSPH, Principal Investigator — Vanderbilt University
Locations (4):
- United States (4):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Orthopaedic Institute, Sioux Falls, South Dakota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided